CLINICAL TRIAL: NCT06714123
Title: Senicapoc in Patients With Progressive Fibrotic ILD (Interstitial Lung Disease) and IPF (Idiopathic Pulmonary Fibrosis) to Prevent Progression.
Brief Title: Senicapoc in Patients With Worsening Fibrotic Interstitial Lung Disease
Acronym: FIBROPOC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Collaborators: Odense Patient Data Explorative Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Fibropoc; 2024-511131-97-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-26; First posted 2024-12-03 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Fibrosis, Interstitial Lung Disease; Idiopathic Pulmonary Fibrosis
Keywords: pulmonary fibrosis; Senicapoc; interstitial lung disease
MeSH Terms: conditions — Pulmonary Fibrosis; Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis | interventions — senicapoc

STUDY DESIGN:
Intervention Model Description: Multicenter, International
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Senicapoc (Active Comparator): Senicapoc 30 mg per day, administered as 3 tablets of 10 mg,.
  Interventions: Drug: Senicapoc
- Placebo (Placebo Comparator): Tablets similar in size, color and composition, as the active comparator, administered as 3 tablets a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Senicapoc — administering 30 mg senicapoc a day, in addition to standard of care.
  Arms: Senicapoc
Drug: Placebo — Tablets similar in size and color
  Arms: Placebo

SUMMARY:
This study will investigate whether the senicapoc drug can prevent the scarring from worsening in interstitial lung disease.

Researchers will compare Senicapoc to a placebo (a look-alike substance that contains no drug) to see if Senicapoc works to prevent lung function worsening.

Participants will be asked to take 3 tablets a day for 26 weeks. Within this period, doctors will follow the participants, ask for experience of adverse events, check lung function and organ status, and participants will need to fill out quality-of-life questionnaires. A total of 5 visits are required, at initiation, after4, 13, 26 and 52 weeks. The final visit will occur 52 weeks after initiation and consist of a normal visit in the outpatient clinic where the doctor asks for relevant information regarding the period after end of administration of the study drug.

DETAILED DESCRIPTION:
Background: Fibrosing interstitial lung disease (F-ILD) represents a heterogeneous group of chronic, severely debilitating, and ultimately lethal lung diseases with limited treatment options. The common denominator for F-ILD is similarities regarding development of scarring of the lungs. Two antifibrotic treatments (pirfenidone, nintedanib), have shown to improve progression free survival, and slowed the decline in forced ventilatory capacity (FVC). These treatments are currently approved in the European Union and are standard of care for many patients. But both treatments have a lot of unbeneficial side-effects, making it unbearable for many patients to receive full dose treatment and often patients progress despite antifibrotic treatment.

Senicapoc is a selective and highly potent inhibitor of KCa3.1 channels. The KCa3.1 channel is pivotal in Ca+ signaling and plays a central role in fibroblast processes. It is therefore thought to play an important role in the development of many fibrotic diseases, including lung fibrosis. Two lines of evidence using human lung cells and lung slices indicate that blocking of the KCa3.1 channel attenuates many profibrotic activities and support the expected antifibrotic effect of senicapoc. In sheep studies, senicapoc has shown not only to attenuate disease progression but also signs of reversing the disease. It has been extensively tested in animal studies and shown no toxic or unbeneficial effects, and it has been tested in human studies in healthy volunteers, patients with sickle cell disease, asthma, and COVID-19, without revealing any serious adverse reactions.

Aims, Objectives and hypothesis: The aim of this study is to investigate the effect of senicapoc in preventing progression in F-ILD. Evaluation will consist of spirometry, 6-minute walking distance test and diffusion capacity. Sidewise changes in quality of life and degree of dyspnea will be obtained. Clinical examinations and bloodtests will be done to evaluate a second aim of this study; the safety of senicapoc in IPF patients.

The hypothesis is that senicapoc is safe, without any major adverse reactions, and has a valuable effect in preventing progression in fibrotic ILD.

Patients diagnosed with fibrotic ILD and shown to progress despite standard of care are candidates. Patients must have an F-ILD diagnosis within 5 years, and an HRCT scan within the previous 24 months. In addition to this, patients must have shown disease progression within the last year, and with no more additional antifibrotic treatment options available. Patients will be recruited from the outpatient clinic. A total of 140 participants will be included, distributed between 6 different sites.

Intervention: Participants will be randomly assigned to one of two groups to receive either senicapoc 30mg/day or placebo in addition to their usual antifibrotic treatment, if any. The tablets containing the active ingredient will have a dosage of 10 mg each, while the placebo tablets are manufactured to resemble the active ingredient tablets in terms of size, color, and design. Participants will be examined at initiation, after 4, 13 and 26 weeks of study drug intake. In addition blood test will be drawn at 0, 4 and 26 weeks. The main trial endpoint is rate of decline of FVC (in mL) over a period of 26 weeks. A final observation will be caried out at week 52, including blood safety assesment.

ELIGIBILITY:
Inclusion Criteria:

* Progressive fibrotic ILD or Progressive IPF diagnosed according to ATS/ERS/JRS/ALAT guidelines at the time of diagnosis
* Age > 18 years
* HRCT historically performed within 24 months
* FVC > 45 %, FEV1/FVC > 0,7 or above LLN
* Annual FVC decline of at least 5% predicted, based on at least three FVC measurements within 6-24 months before enrolment
* Subject able to give informed consent.
* The extent of fibrotic changes is greater than the extent of emphysema on the most recent HRCT scan
* Male subjects of reproductive potential agree to use highly effective contraception/preventive exposure measures from the time of first dose of IMP during the study, and until 90 days (male) after the last dose of IMP.
* Female subjects agree to use highly effective contraceptive during the study, and must show a negative pregnancy test before inclution.
* Able to walk at least 150 meters during the 6MWT at screening Visit 1;
* Able to read and complete the EQ-5D, SGRQ-I, K-BILD questionnaire.

Exclusion Criteria:

* Sickle cell disease
* Any clinical condition or other condition or circumstance that, in the opinion of the investigator, may make a subject unsuitable for inclusion or unlikely or unable to complete the study or comply with study procedures and requirements.
* Known hypersensitivity to any of the IMP ingredients or a history of a significant allergic reaction to any drug as determined by the investigator
* A current immunosuppressive condition
* Clinically significant abnormalities detected on ECG of either rhythm or conduction,
* Moderate to severe hepatic impairment (Child-Pugh B or C); and/or abnormal LFT at screening,
* Clinical laboratory test suggestive of cholestasis with total serum bile acid levels > 3xULN.
* Abnormal renal function, defined as eGFT > 30 ml/kg
* History of malignancy within the past 5 years
* Previous participation in a clinical study with IMP for fibrotic disease within the last 6 months.
* Concurrent participation in another interventional drug, device, or biological investigational research study, or use of an investigational agent within 5 half-lives of the agent
* Lower respiratory tract infection requiring treatment within 4 weeks prior to screening and/or during the screening period.
* History of lung volume reduction surgery or lung transplant.
* Diagnosis of severe pulmonary hypertension
* Unstable cardiovascular, pulmonary (other than IPF), or other disease within 6 months prior to screening or during the screening period
* Use of any of the following therapies within 4 weeks prior to screening and during the screening period, or planned during the study: warfarin, imatinib, ambrisentan, azathioprine, cyclophosphamide, cyclosporine A, bosentan, methotrexate, sildenafil (except for occasional use), prednisone at steady dose > 10 mg/day or equivalent.
* Current alcohol or substance abuse in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The rate of decline of forced vital capacity (FVC) in mL of predicted. | 26 weeks
  Between baseline and 26 weeks

SECONDARY OUTCOMES:
The rate of decline of forced vital capacity (FVC) in % of predicted. | 26 weeks
  Between baseline and 26 weeks.
All cause mortality | 26 weeks
Time to first respiratory-related hospitalization | 26 weeks
Number and degree of adverse events after 26 weeks of treatment. | 26 weeks
  Evaluation of the amount and type of adverse events during the study, and their relation to the study drug
Change in the quality of life after 26 weeks of treatment | 26 weeks
  Measured using specific validated questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Ole Hilberg, Proffesor, Study Director — Sygehus Lillebælt - Vejle
Locations (3):
- Denmark (2):
  - Aarhus University Hospital, Aarhus N
  - Odense University Hospital, Odense C
- Tartu University Hospital,, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: Yes
Procedures, including re-coding of key variables, will be put in place to allow for complete de-identification of the data. All relevant trial-related documents, including the protocol, data dictionary, and the main statistical code, will be made available for sharing along with the data. Data will be completely anonymized according to European law.
  The method for datasharing has yet to be decided.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Six months after the publication of the results, all de-identified individual patient data will be made available for data sharing. There will be no predetermined end-date for the data sharing.
Access Criteria: Data will be available for any research purpose to all interested parties who have approval from an independent review committee and who have a methodological sound proposal as determined by the steering committee of the current trial. Only the methodological qualities and not the purpose or objective of the proposal will be considered. Interested parties will be able to request the data by contacting the principal investigator.